CLINICAL TRIAL: NCT04882618
Title: Is the Extended Lymph Node Dissection Under Indocyanine Green (ICG) Based Fluorescence Imaging Superior to Conventional Extended Lymph Node Dissection During Laparoscopic Radical Prostatectomy(LRRP)?
Brief Title: Use of Indocyanine Green During Pelvic Lymph Node Dissection in Prostate Cancer.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Abdullah Demirtas, MD, Professor in Urology, TC Erciyes University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TSA-2019-9393
Record Dates: First submitted 2021-01-31; First posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Prostate Cancer; Lymph Node Metastases
Keywords: indocyanine green based fluorescence imaging; extendend lymph node dissection; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Lymphatic Metastasis | interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: Prospective single arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICG group (Experimental): ICG injection before LRRP via cystoscopy
  Interventions: Drug: Indocyanine green

INTERVENTIONS:
Drug: Indocyanine green — indocyanine green application during LRRP to detect positive lymph nodes. ICG will be injected to prostate lobes via csytoscopy
  Other Names: Conventional ELND

SUMMARY:
Standard treatment of local or locally advanced prostate cancer is radical prostatectomy (RRP) surgery. During RRP in certain patients extended lymph node dissection (ELND) is recommended. to detect eligible patients for ELND some nomograms based on clinical factors of them is used. The Briganti nomogram is one of them. If the patient has 7% or more probability on Briganti nomogram, then ELND is recommended. But ELND is complicated surgical procedure and may cause labor lost and cost.

It is aimed here to show whether the ICG based fluorescence imaging during laparoscopy may yield higher accuracy to detect metastatic LNs than the conventional ELND?

DETAILED DESCRIPTION:
50 patients with diagnosis of local or locally advance prostate cancer and having LN invasion probability between 7-50% on 2018 Briganti Nomogram will be included to this study.

Before Laparoscopic radical prostatectomy (LRRP), ICG is injected left and right lobe of the propagate during cystoscopy.

Extended LND is performed in all patients. But before it, fluorescence imaging will be done, and ICG positive lymph nodes (LN) are dissected and sent pathology separately.

Positive LN yield pf ICG guided LND and conventional LND is compared.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally limited prostate cancer;
* Intermediate or high risk tumor
* Recommended and planned prostatectomy;
* Completed and signed written consent;
* Voluntarily agreement to participate in this study
* Age of the study participants ≥ 18 years.

Exclusion Criteria:

* Allergic reaction to active ingredient (indocyanine green);
* Iodine allergy;
* Hyperthyroidism;
* High-grade renal impairment;
* High-grade hepatic insufficiency;
* Unwillingness to the storage and disclosure of pseudonymous disease and personal data
* psychiatric pre-existing conditions or other circumstances that make a cooperation by the patient in question

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-11-08 (Actual); Primary Completion 2021-11-08 (Estimated); Study Completion 2021-11-08 (Estimated)

PRIMARY OUTCOMES:
Indocyanine green postive lymph node numbers | 15 day after surgery
  total number of dissected lymph nodes which are indocyanine green positive
Total lymph node numbers of conventional extended lymph node dissection | 15 day after surgery
  total number of dissected lymph nodes during conventional extended lymph node dissection
pathology of indocyanine green positive lymph nodes | 15 day after surgery
  İndocyanine green positvie lymph nodes are malign or benign
pathology of lymph nodes | 15 day after surgery
  Pathology of material from conventional extended lymph node dissection

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah A Demirtaş, Md, Prof, Principal Investigator — TC Erciyes University
Locations (1):
- Department of Urology, Ercieys University, Faculty Of Medicine,, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No